CLINICAL TRIAL: NCT00000213
Title: IV Cocaine Abuse: A Laboratory Model
Brief Title: IV Cocaine Abuse: A Laboratory Model - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-06234-2; R01DA006234 (NIH); R01-06234-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2012-12

CONDITIONS: Cocaine-Related Disorders
Keywords: intravenous abuse
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine

SUMMARY:
The purpose of this study is to evaluate the effects of fluoxetine maintenance on cocaine taking and on the physiological and subjective effects of cocaine, including cocaine craving.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1990-04; Primary Completion 1991-04 (Actual); Study Completion 1991-04 (Actual)

PRIMARY OUTCOMES:
Direct cocaine effects
Interaction of cocaine/fluox. on cardio measures
Interaction of cocaine/fluox. on coc's subjective
Effects of fluoxetine on cocaine craving
Drug use during outpatient fluoxetine maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Richard Foltin, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States